CLINICAL TRIAL: NCT04970368
Title: Randomized Phase 3 Study of Selective Versus Sentinel Node Surgical Staging for the Treatment of Endometrial Cancer
Brief Title: Comparison of Nodal Staging in Endometrial Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Frederick R. Ueland, M.D. (Other)
Responsible Party: Sponsor-Investigator, Frederick R. Ueland, M.D., Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21-GYN-210
Record Dates: First submitted 2021-06-25; First posted 2021-07-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Endometrial Cancer
Keywords: Sentinel node; Cancer; Endometrial; Intraoperative Consultation
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sentinel Node Surgical Staging (Experimental)
  Interventions: Procedure: Sentinel node procedure
- Selective Surgical Staging (Experimental)
  Interventions: Procedure: Selective staging

INTERVENTIONS:
Procedure: Sentinel node procedure — Excision of ALL mapped nodes and other suspicious nodes regardless of mapping and label by anatomic location
  Arms: Sentinel Node Surgical Staging
Procedure: Selective staging — Intraoperative consultation (IOC)
  Arms: Selective Surgical Staging

SUMMARY:
This study aims to estimate the recurrence-free survival rates in women with endometrial cancer treated with selective versus sentinel node surgical staging.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for complete hysterectomy and bilateral salpingooophorectomy with pelvic and aortic lymphadenectomy
* Histologically or cytologically confirmed endometrioid-type endometrial cancer confined to the uterine corpus
* No clinical evidence of extra-uterine disease on pre-operative evaluation.
* Prior systemic chemotherapy is allowed so long as it was at least five years prior to study enrollment, and there is no evidence of disease after such therapy.
* Age ≥18 years.
* Life expectancy (estimated survival) of at least 6 months.
* AST(SGOT)/ALT(SGPT) < 3.0X upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* GOG/ECOG Performance Status greater than 2
* Non-endometrioid cell type
* Clinical evidence of disease that extends beyond the uterus, including the presence of suspicious aortic or inguinal nodes on imaging or clinical exam
* Previous vaginal, pelvic or abdominal irradiation
* Chemotherapy, hormone therapy or immunotherapy directed at the present disease
* Previous pelvic lymphadenectomy or retroperitoneal surgery
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Known allergy to iodine or indigocyanine green (ICG) tracer, or allergic reactions to compounds of similar chemical or biologic composition
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival rate | 5 years
  Recurrence-free survival rate in women with endometrial cancer treated with selective versus sentinel node surgical staging

SECONDARY OUTCOMES:
Progression-free survival rate | 5 years
  Progress-free survival rate in women with endometrial cancer treated with selective versus sentinel node surgical staging
Disease-specific survival rate | 5 years
  Disease-specific survival rate in women with endometrial cancer treated with selective versus sentinel node surgical staging
Overall patient survival rate | 5 years
  Overall survival rate in women with endometrial cancer treated with selective versus sentinel node surgical staging
Concordance of SELECTIVE and SENTINEL NODE surgical staging with final pathology | 5 years
  Percentage of participants for whom selective surgical staging and final pathology match. Match incorporates grade, lesion size, depth of invasion, and low-risk (no lymphadenectomy) versus high-risk (lymphadenectomy).
Patient morbidity | 5 years
Patient mortality | 5 years

OTHER OUTCOMES:
Location patterns of nodal involvement associated with staging procedures | 5 years
  Location patterns related to nodal involvement with staging procedures will be reported.
Number of metastatic lymph node(s) associated with staging procedures | 5 years
  The number of metastatic lymph node(s) associated with the staging procedures will be reported.
Patterns of nodal involvement associated with primary tumor grade | 5 years
  Primary tumor grade related to nodal involvement will be reported
Patterns of nodal involvement associated with primary tumor lesion size | 5 years
  Primary tumor lesion size related to nodal involvement will be reported.
Patterns of nodal involvement associated with primary tumor depth of invasion | 5 years
  Primary tumor depth related to nodal involvement will be reported.
Patterns of nodal involvement associated with primary tumor cell type | 5 years
  Primary tumor cell type related to nodal involvement will be reported.
Location patterns of nodal involvement associated with disease stage | 5 years
  Location related to nodal involvement with disease stage will be reported.
Number of metastatic lymph node(s) associated with disease stage | 5 years
  The number of metastatic lymph node(s) associated with the staging procedures will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Ueland, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No